CLINICAL TRIAL: NCT02207062
Title: A Pilot Study of Single-Agent Ibrutinib in Relapsed or Refractory Transformed Indolent B-Cell Non-Hodgkin Lymphoma
Brief Title: Ibrutinib in Treating Patients With Relapsed or Refractory Transformed Indolent B-cell Non-Hodgkin Lymphoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: Janssen Pharmaceuticals (Industry)
Responsible Party: Principal Investigator, Ajay Gopal, Professor, University of Washington
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 9107; NCI-2014-01573 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 9107 (Other: Fred Hutch/University of Washington Cancer Consortium); RG1714041 (Other: Fred Hutch/University of Washington Cancer Consortium)
Record Dates: First submitted 2014-07-30; First posted 2014-08-01 (Estimated); Results first posted 2025-01-07 (Actual); Last update posted 2025-01-07 (Actual); Status verified 2024-11

CONDITIONS: Recurrent Transformed B-Cell Non-Hodgkin Lymphoma; Refractory Transformed B-Cell Non-Hodgkin Lymphoma
Keywords: Non-Hodgkin Lymphoma
MeSH Terms: conditions — Lymphoma, Non-Hodgkin | interventions — ibrutinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Treatment (ibrutinib) (Experimental): Patients receive ibrutinib PO QD in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Ibrutinib; Other: Laboratory Biomarker Analysis

INTERVENTIONS:
Drug: Ibrutinib — Given PO
  Other Names: BTK Inhibitor PCI-32765; CRA-032765; PCI-32765
Other: Laboratory Biomarker Analysis — Correlative studies

SUMMARY:
This pilot phase II trial studies ibrutinib in treating patients with transformed indolent (a type of cancer that grows slowly) B-cell non-Hodgkin lymphoma that have returned after a period of improvement (relapsed) or do not respond to treatment (refractory). Ibrutinib may stop the growth of cancer cells by blocking some of the enzymes (proteins) needed for cell growth.

DETAILED DESCRIPTION:
OUTLINE:

Patients receive ibrutinib orally (PO) once daily (QD) in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up every 3 months for up to 5 years.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically confirmed transformed indolent B-cell non-Hodgkin lymphoma that is relapsed or refractory to at least one line of therapy
* Patients must have a computed tomography (CT) (preferred) or magnetic resonance imaging (MRI) scan of the chest, abdomen, and pelvis within 28 days of enrollment
* Patients must have measurable disease defined as lesions greater than 1.5 cm that can be accurately measured in two dimensions by CT (preferred), or MRI
* Patients must have a positron emission tomography (PET) scan within 56 days of enrollment
* Patients must have an Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 2
* Absolute neutrophil count (ANC) >= 1000/mm^3 or >= 750/mm^3 in the setting of marrow involvement by disease
* Platelets >= 50,000/mm^3 or >= 30,000/mm^3 in the setting of marrow involvement by disease or splenomegaly due to disease
* Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) =< 3 x upper limit of normal (ULN)
* Total bilirubin =< 1.5 x ULN unless bilirubin rise is due to Gilbert's syndrome or of non-hepatic origin
* Creatinine clearance (Clcr) > 25 mL/min
* Patients must be anticipated to complete 2 cycles of therapy in the opinion of the treating physician
* Women of childbearing potential and men who are sexually active must affirm they are practicing a highly effective method of birth control during and after the study consistent with local regulations regarding the use of birth control methods for subjects participating in clinical trials; men must agree to not donate sperm during or after the study; for females, these restrictions apply for 1 month after the last dose of study drug; for males, these restrictions apply for 3 months after the last dose of the study drug
* Women of childbearing potential must have a negative serum (beta-human chorionic gonadotropin [beta-hCG]) or urine pregnancy test at screening; women who are pregnant or breastfeeding are ineligible for this study
* Sign (or their legally-acceptable representatives must sign) an informed consent document in accordance with institutional and federal guidelines indicating that they understand the investigational nature of and procedures required for the study, including biomarkers, and are willing to participate in and comply with the guidelines of the study

Exclusion Criteria:

* Known history of human immunodeficiency virus (HIV) or active hepatitis C virus or active hepatitis B virus infection or any uncontrolled active systemic infection
* Major surgery or a wound that has not fully healed within 4 weeks of initiation of therapy
* Known central nervous system lymphoma
* History of stroke or intracranial hemorrhage within 6 months of screening
* Requires anticoagulation with warfarin or equivalent vitamin K antagonists (e.g., phenprocoumon)
* Requires chronic treatment with strong cytochrome P450, family 3, subfamily A (CYP3A) inhibitors
* Clinically significant cardiovascular disease such as uncontrolled or symptomatic arrhythmias, congestive heart failure, or myocardial infarction within 6 months of screening, or any class 3 (moderate) or class 4 (severe) cardiac disease as defined by the New York Heart Association Functional Classification
* Vaccinated with live, attenuated vaccines within 4 weeks of initiation of therapy
* Any life-threatening illness, medical condition, or organ system dysfunction which, in the investigator's opinion, could compromise the subject's safety, interfere with the absorption or metabolism of ibrutinib capsules, or put the study outcomes at undue risk
* Patients with other prior malignancies except for adequately treated basal cell carcinoma, squamous cell carcinoma of the skin, breast or cervical cancer in situ, or other cancer from which the patient has been disease-free for 5 years or greater, unless approved by the protocol sponsor-investigator/lead-sub-investigator
* Patients that previously were treated with ibrutinib for > 7 days
* Previous chemotherapy, immunotherapy, biologically targeted therapy, other investigational agent, or radiation therapy within 3 weeks of initiation of ibrutinib therapy or radio-immunotherapy within 12 weeks of initiation of ibrutinib therapy
* Prior allogeneic transplant with graft-versus-host disease (GVHD) requiring immunosuppressive therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2014-10; Primary Completion 2023-11-01 (Actual); Study Completion 2023-11-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ajay K. Gopal, Principal Investigator — Fred Hutch/University of Washington Cancer Consortium
Locations (1):
- Fred Hutch/University of Washington Cancer Consortium, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Treatment (Ibrutinib)
Started | 20
Completed | 20
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Treatment (Ibrutinib)
Number analyzed (Participants) | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 8
  >=65 years | 12
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11
  Male | 9
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 18
  Unknown or Not Reported | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 18
  More than one race | 0
  Unknown or Not Reported | 1
Region of Enrollment [Number; unit: participants]
  United States | 20

OUTCOME MEASURES:

1. Primary Outcome: Overall Response Rate (Combined Complete Response + Partial Response)
Time Frame: Up to 5 years
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Ibrutinib)
Number analyzed (Participants) | 18
Participants | 6

2. Secondary Outcome: Complete Response Rate
Time Frame: Up to 5 years
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Ibrutinib)
Number analyzed (Participants) | 18
Participants | 2

3. Secondary Outcome: Disease Control Rate
Time Frame: >12 months
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Ibrutinib)
Number analyzed (Participants) | 20
Participants | 4

4. Secondary Outcome: Overall Survival
Time Frame: Up to 5 years
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Treatment (Ibrutinib)
Number analyzed (Participants) | 20
months | 22.4 [7.5 to 36.4]

5. Secondary Outcome: Progression-free Survival
Description: Progression-free survival will be calculated using assessments by investigators. Kaplan-Meier methodology will be used to estimate event-free curves and corresponding quartiles (including the median).
Time Frame: Time from first study drug administration to the first occurrence of disease progression or death from any cause, assessed up to 5 years
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Treatment (Ibrutinib)
Number analyzed (Participants) | 20
months | 4.1 [2.4 to 6.2]

6. Secondary Outcome: Response Rate Relative to the Underlying B-cell Histology
Description: Participants with a histology of follicular lymphoma at diagnosis achieving at least a partial response to treatment.
Time Frame: Up to 5 years
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Ibrutinib)
Number analyzed (Participants) | 18
Participants | 4

7. Secondary Outcome: Tolerability of Chronic Ibrutinib Therapy
Description: The National Cancer Institute Common Terminology Criteria for Adverse Events version 4.0 will be used to classify and grade toxicities. Count of participants who stopped ibrutinib due to toxicities.
Time Frame: Up to 5 years
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Ibrutinib)
Number analyzed (Participants) | 20
Participants | 1

ADVERSE EVENTS:
Time Frame: Adverse events will be collected from the time the consent is signed until 30 days following the last dose of study drug, an average of 18 months. All-Cause Mortality assessed up to 5 years.
Arm/Group | Treatment (Ibrutinib)
All-Cause Mortality (participants affected / at risk) | 14/20
Serious Adverse Events (participants affected / at risk) | 7/20
Other Adverse Events (participants affected / at risk) | 20/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Ibrutinib) (N=20)
Nausea (Gastrointestinal disorders) | 1 (1)
Pericarditis (Cardiac disorders) | 1 (1)
Atrial Fibrillation (Cardiac disorders) | 2 (2)
Groin Pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) — Pain in right hip
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Mucositis (Gastrointestinal disorders) | 1 (1)
Esophagitis (Gastrointestinal disorders) | 1 (1)
Pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Acute Myocardial Infarction (Cardiac disorders) | 2 (2)
Sepsis (Infections and infestations) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1)
Abdominal Pain (Gastrointestinal disorders) | 1 (1) — Right lower quandrant
Flu-like symptoms (Infections and infestations) | 1 (1)
Clamminess (General disorders) | 1 (1)
Fatigue (General disorders) | 1 (1)
Ventricular arrythmia (Cardiac disorders) | 1 (1)
CHF Exacerbation (Cardiac disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Ibrutinib) (N=20)
Alanine aminotransferase increased (Investigations) | 3 (6)
Anorexia (Metabolism and nutrition disorders) | 2 (3)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (2)
Aspartate aminotransferase increased (Investigations) | 2 (2)
Atrial Fibrillation (Cardiac disorders) | 3 (4)
Back Pain (Musculoskeletal and connective tissue disorders) | 2 (2)
Bruising (Injury, poisoning and procedural complications) | 12 (13)
Constipation (Gastrointestinal disorders) | 4 (5)
Cough (Respiratory, thoracic and mediastinal disorders) | 3 (6)
Diarrhea (Gastrointestinal disorders) | 6 (7)
Dizziness (Nervous system disorders) | 3 (3)
Dry Mouth (Gastrointestinal disorders) | 2 (3)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Edema Limbs (General disorders) | 4 (7)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 3 (5)
Esophagitis (Gastrointestinal disorders) | 2 (5)
Fatigue (General disorders) | 11 (12)
Fever (General disorders) | 2 (3)
Loose Stools (Gastrointestinal disorders) | 2 (3)
Cold-Like Symptoms (Infections and infestations) | 2 (3)
Headache (Nervous system disorders) | 2 (2)
Hypertension (Vascular disorders) | 3 (3)
Hypokalemia (Metabolism and nutrition disorders) | 2 (2)
Mucositis oral (Gastrointestinal disorders) | 2 (4)
Nausea (Gastrointestinal disorders) | 4 (5)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3 (3)
Peripheral sensory neuropathy (Nervous system disorders) | 2 (2)
Pruritus (Skin and subcutaneous tissue disorders) | 2 (2)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 3 (5)
Bronchitis (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Brittle nails (Skin and subcutaneous tissue disorders) | 3 (3)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Upper respiratory infection (Infections and infestations) | 2 (2)
Urinary urgency (Renal and urinary disorders) | 2 (2)
Vomiting (Gastrointestinal disorders) | 4 (6)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-06-28): https://cdn.clinicaltrials.gov/large-docs/62/NCT02207062/Prot_SAP_000.pdf